CLINICAL TRIAL: NCT04792788
Title: The Use of Neurally Adjusted Ventilator Assist Versus Pressure Support Ventilation durIng weaninG From Mechanical ventilAtion in pediaTric Patients After livEr Transplantation. A Physiologic Cross-over Controlled Trial. NAVIGATE Study
Brief Title: NAVA vs PSV Ventilation During Weaning From Mechanical Ventilation in Children After Liver Transplantation
Acronym: NAVIGATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1695_OPBG_2018
Record Dates: First submitted 2021-02-03; First posted 2021-03-11 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Liver Transplantation; Weaning From Mechanical Ventilation
Keywords: mechanical ventilation; liver transplantation; pediatric; neurally adjusted ventilatory assist; weaning; pressure support ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAVA/PSV/NAVA (Active Comparator): 6 patients
  Interventions: Procedure: Weaning from mechanical ventilation
- PSV/NAVA/PSV (Active Comparator): 6 patients
  Interventions: Procedure: Weaning from mechanical ventilation

INTERVENTIONS:
Procedure: Weaning from mechanical ventilation — Cross over study: 3 periods of 40 minutes in ventilation mode (NAVA or PSV); to register ventilator traces and cardiopulmonary parameters during the last 10 minutes of each period.

SUMMARY:
Liver transplantation is the treatment of choice for acute and chronic end-stage liver disease. Neurally Adjusted Ventilator Assist (NAVA) may be a feasible solution to guide the liberation from mechanical ventilation reducing asynchronies between patient and ventilator, and optimizing ventilator cycling. Cardiovascular and respiratory effects during NAVA ventilation are very limited after major abdominal surgery. The purpose of this application is to explore the efficacy of NAVA to reduce the asynchronies between the ventilator and pediatric patient admitted in Pediatric Intensive Care Unit (PICU) after major abdominal surgery, and the relationship between an optimal level of NAVA and cardiac and pulmonary function.

DETAILED DESCRIPTION:
Twelve pediatric patients underwent liver transplantation and admitted during postoperative period in PICU will be studied. They will be endotracheally intubated and spontaneously triggering the mechanical ventilator. In each patient enrolled a specially manufactured nasogastric tube will be inserted. This nasogastric tube is equipped with ten electrodes. The correct position of the nasogastric tube (and of electrodes) will be confirmed checking the good quality of Edi trace with the P waves displayed by the central electrodes on monitor of Servo I Ventilator (Maquet). All the patients will be ventilated using ventilators with NAVA option (Servo-I, Maquet Critical Care, Sweden). After a stabilization period in Pressure Support Ventilation (PSV) according with the attending physician, each patient will be studied for a duration of 2 hours, divided in three trials of 40-minutes (first 30 minutes to washout from the effects of previous ventilation mode and during the last 10 minutes the results will be recorded). Each patient will be randomized for ventilation mode sequence (PSV/NAVA/PSV or NAVA/PSV/NAVA). The patient tracings of flow, airway pressure, electrical activity of diaphragm for the patient-ventilator interaction analysis, blood gas analysis and cardiovascular parameters will be recorded during each trial.

ELIGIBILITY:
Inclusion Criteria:

* Liver recipients (from cadaveric or living donor)
* Invasive Mechanical ventilation

Exclusion Criteria:

* Neurological impairment
* Neuromuscular, mitochondrial, metabolic, or chromosomal diseases with baby hypotonia
* Lesions of medulla
* Hemodynamic instability requiring inotropes/vasopressors (dopamine > 6 mcg/kg/min, norepinephrine, epinephrine, dobutamine, milrinone) or volume load.
* Congenital cardiovascular disease
* Patient extubated
* Need of controlled mechanical ventilation
* Intravenous infusion of benzodiazepines or propofol
* Pneumonia, pneumothorax, massive pleural effusion
* Patient placed on extracorporeal circuit
* Contraindications to insert nasogastric tube
* Not expected to survive beyond 24 hours
* Parental/legal guardian refusal

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Asynchrony Index | last 10 minutes of each ventilatory trial, NAVA or PSV
  Asynchrony Index (ratio between the number of asynchronous breathing events and the total respiratory rate, expressed as percentage) will be measured in the last 10 minutes of each ventilatory trial of 40 minutes.
Left and right ventricle function | last 10 minutes of each ventilatory trial, NAVA or PSV
  Evaluation of left and right ventricular function variation during each ventilation mode. It will be measured by trans-thoracic echocardiogram in the last 10 minutes of each ventilatory trial of 40 minutes.

SECONDARY OUTCOMES:
arterial partial pressure of oxygen (PaO2) | last 10 minutes of each ventilatory trial, NAVA or PSV
  millimeters of mercury (mm Hg)
arterial partial pressure of carbon dioxide | last 10 minutes of each ventilatory trial, NAVA or PSV
  mm Hg
oxygen index | last 10 minutes of each ventilatory trial, NAVA or PSV
  {[mean airway pressure in centimeters of water × fraction of inspired oxygen × 100] ÷ PaO2 in mm Hg}
respiratory rate | last 10 minutes of each ventilatory trial, NAVA or PSV
  breaths per minute
lactate | last 10 minutes of each ventilatory trial, NAVA or PSV
  millimole/liter
heart rate | last 10 minutes of each ventilatory trial, NAVA or PSV
  beats per minute (bpm)
cardiac index | last 10 minutes of each ventilatory trial, NAVA or PSV
  {cardiac output [stroke volume (milliliter) x heart rate (bpm)] / body surface area (BSA; weight in kilograms and height in centimeters will be combined to report BSA in m^2)} in liters/minute/m^2
mean arterial pressure | last 10 minutes of each ventilatory trial, NAVA or PSV
  mm Hg
central venous pressure | last 10 minutes of each ventilatory trial, NAVA or PSV
  mm Hg
systemic vascular resistance | last 10 minutes of each ventilatory trial, NAVA or PSV
  [(mean arterial pressure - central venous pressure) x 79.92 / cardiac index] in dynes/seconds/cm^-5

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Chiusolo, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Fabrizio Chiusolo, Rome, RM, Italy

REFERENCES:
- [Background] Esquivel CO, Iwatsuki S, Gordon RD, Marsh WW Jr, Koneru B, Makowka L, Tzakis AG, Todo S, Starzl TE. Indications for pediatric liver transplantation. J Pediatr. 1987 Dec;111(6 Pt 2):1039-45. doi: 10.1016/s0022-3476(87)80053-7. PMID 3316578
- [Background] Ulukaya S, Arikan C, Aydogdu S, Ayanoglu HO, Tokat Y. Immediate tracheal extubation of pediatric liver transplant recipients in the operating room. Pediatr Transplant. 2003 Oct;7(5):381-4. doi: 10.1034/j.1399-3046.2003.00072.x. PMID 14738299
- [Background] Fullington NM, Cauley RP, Potanos KM, O'Melia L, Zurakowski D, Bae Kim H, Seefelder C, Vakili K. Immediate extubation after pediatric liver transplantation: a single-center experience. Liver Transpl. 2015 Jan;21(1):57-62. doi: 10.1002/lt.24036. PMID 25368908
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Background] Coisel Y, Chanques G, Jung B, Constantin JM, Capdevila X, Matecki S, Grasso S, Jaber S. Neurally adjusted ventilatory assist in critically ill postoperative patients: a crossover randomized study. Anesthesiology. 2010 Oct;113(4):925-35. doi: 10.1097/ALN.0b013e3181ee2ef1. PMID 20823760
- [Background] Antonelli M, Conti G, Bufi M, Costa MG, Lappa A, Rocco M, Gasparetto A, Meduri GU. Noninvasive ventilation for treatment of acute respiratory failure in patients undergoing solid organ transplantation: a randomized trial. JAMA. 2000 Jan 12;283(2):235-41. doi: 10.1001/jama.283.2.235. PMID 10634340
- [Background] Moulin D, Clement de Clety S, Reynaert M, Carlier MA, Veyckmans F, Claus D, Buts JP, de Hemptinne B, Otte JB. Intensive care for children after orthotopic liver transplantation. Intensive Care Med. 1989;15 Suppl 1:S71-2. doi: 10.1007/BF00260893. PMID 2656816
- [Background] Chidini G, De Luca D, Conti G, Pelosi P, Nava S, Calderini E. Early Noninvasive Neurally Adjusted Ventilatory Assist Versus Noninvasive Flow-Triggered Pressure Support Ventilation in Pediatric Acute Respiratory Failure: A Physiologic Randomized Controlled Trial. Pediatr Crit Care Med. 2016 Nov;17(11):e487-e495. doi: 10.1097/PCC.0000000000000947. PMID 27749511
- [Background] Scharf SM, Caldini P, Ingram RH Jr. Cardiovascular effects of increasing airway pressure in the dog. Am J Physiol. 1977 Jan;232(1):H35-43. doi: 10.1152/ajpheart.1977.232.1.H35. PMID 319686
- [Background] Vieillard-Baron A, Loubieres Y, Schmitt JM, Page B, Dubourg O, Jardin F. Cyclic changes in right ventricular output impedance during mechanical ventilation. J Appl Physiol (1985). 1999 Nov;87(5):1644-50. doi: 10.1152/jappl.1999.87.5.1644. PMID 10562603
- [Derived] Chiusolo F, Spinazzola G, Costa R, Franceschini A, Tortora F, Polisca F, Rossetti E, Rava L, Chinali M, Fanelli V, Conti G. Effect of neurally adjusted ventilator assist versus pressure support ventilation on asynchronies and cardiac function in pediatric liver transplantation. Sci Rep. 2025 Feb 28;15(1):7158. doi: 10.1038/s41598-025-91590-z. PMID 40021754